CLINICAL TRIAL: NCT03060642
Title: Application of the Microbiome and Microenvironment to Novel Non-Endoscopic Screening and Surveillance in Barrett's Esophagus
Brief Title: The Microenvironment in Barrett's Esophagus
Acronym: BETRNet2
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Mayo Clinic (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Julian A Abrams, MD, Assistant Professor of Medicine and Epidemiology, Columbia University
Other Study IDs: AAAQ8763; NCI U54 CA163004-09 (Other: National Cancer Institute/NIH/ DHHS)
Record Dates: First submitted 2017-02-02; First posted 2017-02-23 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
Keywords: Microenvironment; Microbiome; Screening; Barrett Esophagus; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva Gastric Aspirate Tissue from the Esophagus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Barrett's esophagus: Barrett's esophagus, without or with dysplasia or adenocarcnoma
  Interventions: Device: Tethered capsule sponge; Device: Electronic nose device
- Controls: Non-BE endoscopic controls
  Interventions: Device: Tethered capsule sponge; Device: Electronic nose device

INTERVENTIONS:
Device: Tethered capsule sponge — Subjects swallow a tethered capsule sponge sampling device, which is then withdrawn through the mouth after an interval of 5 minutes.
  Other Names: EsophaCap
Device: Electronic nose device — Subjects breathe into the device, which then records an exhaled volatile organic compounds (VOC) signature.
  Other Names: Aeonose

SUMMARY:
This study aims to elucidate the relationship between the microbiome, inflammation, and the microenvironment in Barrett's esophagus (BE) and esophageal adenocarcinoma (EAC), with the end goal of developing a non-endoscopic testing strategy based on pathogenic factors to identify patients at highest risk for EAC. To accomplish this the investigators will enroll 100 patients with known BE (50 with dysplasia or EAC) and 50 subjects without BE undergoing upper endoscopy. Prior to endoscopy each subject will undergo three minimally invasive potential screening and surveillance tests: saliva (oral microbiome), breath test (exhaled volatile organic compounds), and tethered capsule sponge sampling (methylated DNA markers). The study will evaluate these novel tests in combination with clinical and anthropometric factors to describe an optimal strategy for BE screening and monitoring.

DETAILED DESCRIPTION:
The investigators will perform a multi-center cross-sectional study of patients with Barrett's esophagus, with and without associated dysplasia or cancer, and controls without BE. Enrollment of controls will be stratified based on use of proton pump inhibitors (PPIs). The investigators plan to enroll an approximate total of 150 subjects:

100 BE patients (with or without associated dysplasia or cancer)

* 50 subjects with non-dysplastic BE
* 50 subjects with BE and dysplasia or EAC

  50 controls
* 25 controls on PPIs (at least once daily)
* 25 controls not taking PPIs

Various tests will be performed and samples collected on the day of endoscopy. These tests include: saliva samples, electronic nose device testing, tethered capsule sponge testing, dietary questionnaires, and collection of blood and gastrointestinal biosamples. Analyses of this data and samples will then be performed to address the specific aims above.

ELIGIBILITY:
Inclusion Criteria:

(for BE patients)

* History of histologically confirmed BE, defined as endoscopically-suspected BE with intestinal metaplasia with goblet cells on esophageal biopsies
* BE length M≥2
* Taking proton pump inhibitors at least once daily for 3 months prior to enrollment
* Age ≥18

Exclusion Criteria:

* History of gastric cancer or esophageal squamous cell cancer
* History of gastric or esophageal surgery
* Use of antibiotics or systemic immunosuppressants within three months prior to the date of endoscopy (intranasal and inhaled steroids are allowed)
* Known untreated esophageal stricture or uninvestigated dysphagia
* Inability to give informed consent
* (BE patients only) History of prior endoscopic therapy for BE except a history of prior endoscopic mucosal resection (EMR) of focal lesions without subsequent ablative therapy is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without Barrett's esophagus already scheduled for upper endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Oral and esophageal 16S rRNA gene sequencing | 1 day
  Oral and esophageal microbiome

SECONDARY OUTCOMES:
Esophageal tissue RNA-Seq | 1 day
  Esophageal tissue transcriptome
Gastric aspirate mass spectrometry | 1 day
  Gastric aspirate bile acid composition

CONTACTS AND LOCATIONS:
Overall Officials: Julian A. Abrams, MD, MS, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Iyer PG, Slettedahl SW, Mahoney DW, Giakoumopoulos M, Olson MC, Krockenberger M, Taylor WR, Foote P, Berger C, Leggett C, Wu TT, Antpack E, Falk GW, Ginsberg GG, Abrams JA, Lightdale CJ, Ramirez F, Kahn A, Wolfsen H, Konda V, Trindade AJ, Kisiel JB. Algorithm Training and Testing for a Nonendoscopic Barrett's Esophagus Detection Test in Prospective Multicenter Cohorts. Clin Gastroenterol Hepatol. 2024 Aug;22(8):1596-1604.e4. doi: 10.1016/j.cgh.2024.03.003. Epub 2024 Mar 19. PMID 38513982